CLINICAL TRIAL: NCT06960226
Title: Reducing Pain Thresholds Using a Focused Music Listening Technique
Brief Title: Replication Study: Reducing Pain With Focused Music Listening
Acronym: PainMusic2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Collaborators: The Research Council of Norway (Other); European Research Council (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REK NR 2019/1031 7236
Record Dates: First submitted 2025-04-28; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Pain; Pain Management; Pain Threshold; Painful; Pain Intensity; Pain Intervention; Psychomotor Performance; Healthy Volunteers
Keywords: Pain; Pain Perception; Experimental Pain; Analgesia; Music; Music Listening; Sensorimotor Synchronization; Tapping; Rhythm; Electrical Pain Stimulation; Replication Study; Endogenous Opioid System; Attention; Emotion; Affect; Pain Management; Music Therapy
MeSH Terms: conditions — Pain; Agnosia

STUDY DESIGN:
Intervention Model Description: All participants experience all conditions within a 2x2 within-subjects factorial design. Factors crossed are: 1. Auditory Condition (Music versus Silence) and 2. Task Condition (Active Sensorimotor Synchronization versus Passive Control). The Active task involves participants synchronizing movements (e.g., foot tapping, head nodding) to music or a pacing stimulus. The Passive task requires participants to remain still without performing these specific movements. This results in four experimental conditions: Music+Active, Music+Passive (Listening only), Silence+Active, and Silence+Passive. The order of these conditions is counterbalanced across participants. Brief, non-invasive electrical pain stimuli are delivered to the forearm during experimental trials.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Within-Subjects Conditions (Experimental): All participants experience all conditions in a 2x2 within-subjects factorial design. Interventions manipulate two factors: 1. Auditory Condition: Participants listen to selected music (via headphones) or experience silence. 2. Task Condition: Participants perform Active Sensorimotor Synchronization (syncing foot taps/head nods to music or pacing stimulus) or maintain Passive Control (remaining still). Each participant completes trials for all 4 resulting conditions: Music+Active, Music+Passive, Silence+Active, Silence+Passive. Condition order is counterbalanced across participants. During trials, brief non-invasive electrical pain stimuli (BIOPAC system) are delivered to the forearm; intensity is individually calibrated based on pain threshold. Key outcomes (perceived pain, emotional state ratings) are collected.
  Interventions: Other: Music Listening; Other: Silence Control; Other: Active Sensorimotor Synchronization; Other: Passive Control Task

INTERVENTIONS:
Other: Music Listening — Participants listen to selected instrumental music excerpts presented via headphones during designated experimental trials.
Other: Silence Control — Participants experience periods of silence with no music presented via headphones during designated control trials. This serves as the auditory control condition compared to Music Listening.
Other: Active Sensorimotor Synchronization — Participants actively synchronize movements (such as foot tapping and/or head nodding) by timing them with the rhythm of the presented music or with a pacing stimulus provided during silent trials.
Other: Passive Control Task — Participants remain still and do not perform specific instructed synchronized movements during designated control trials. This serves as the motor task control condition compared to Active Sensorimotor Synchronization.

SUMMARY:
The goal of this clinical trial is to confirm previous findings that actively tapping along to music can reduce pain more than just listening to music. This study aims to replicate the findings of a previous study (NCT05267795), with one change in how mild pain is created for the experiment. This study involves healthy adults.

The main questions the study aims to answer are:

1. Does actively tapping along to music lower feelings of pain compared to just listening to music?
2. Does actively tapping along to music lower feelings of pain compared to being in silence (with or without tapping)?
3. Is this method of using music and tapping helpful for managing pain?

Researchers will compare the amount of pain participants feel in four different situations:

1. Listening to music while actively tapping their foot along with it.
2. Just listening to music while resting their foot.
3. Actively tapping their foot in silence.
4. Sitting in silence while resting their foot.

Participants in this study will:

Experience brief moments of mild pain on their forearm. This pain is safely created using a small electrical pulse from a device held gently on the skin by the researcher. (This replaces the pressure method used in the original study).

Sometimes listen to music through headphones, and sometimes sit in silence. Sometimes tap their foot along to the music or a beat, and sometimes rest their foot. Rate how much pain they feel on a number scale after each pain pulse. Answer short questions about their mood during the experiment. Answer questions about how familiar they are with the music and how much they liked it at the end.

DETAILED DESCRIPTION:
This study is a pre-registered replication of a previous trial (NCT05267795) investigating the analgesic effects of sensorimotor synchronization to music. While music listening alone has shown small, albeit reliable, pain-reducing effects, recent theories propose that active synchronization (like tapping or dancing) engages the endogenous opioid system (EOS), potentially leading to stronger analgesia and enhanced social bonding. The original study provided initial evidence supporting this, finding that actively tapping to music significantly reduced experimentally induced pain compared to passive music listening or silence conditions.

This replication study aims to confirm the primary finding that sensorimotor synchronization to music significantly reduces pain perception compared to passive music listening and control conditions. The study employs a 2x2 within-subjects factorial design with two factors: Auditory Condition (Music vs. Silence) and Task Condition (Active Tapping vs. Passive Control). Healthy adult participants will undergo all four conditions.

The primary methodological difference from the original study is the method of pain induction. Instead of pressure algometry, this study will use non-invasive transcutaneous electrical stimulation applied to the participant's forearm via a BIOPAC HSTM01 certified stimulus device. This change was implemented to allow for potentially greater precision and control over the stimulus intensity compared to manual pressure application. Pain intensity will be individually calibrated for each participant based on their pain threshold, ensuring only mild to moderate pain levels are experienced. Safety protocols, including screening for contraindications (e.g., pacemakers, epilepsy, pregnancy, local malignancies) and continuous monitoring, are in place.

Consistent with the original study, perceived pain intensity will be the primary outcome measure, rated on a numerical scale after each stimulus. Secondary measures, including ratings of emotional state (pleasantness, arousal), music familiarity, and music preference, will be collected to explore potential attentional and emotional mechanisms underlying the observed effects, as suggested by the original research. This replication seeks to provide robust evidence regarding the potential for active musical engagement, specifically sensorimotor synchronization, as a tool for pain management.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Self-reported good general health
* Able to understand study procedures and provide informed consent
* Normal or corrected-to-normal hearing (sufficient for music perception)

Exclusion Criteria:

* Contraindications for Electrical Stimulation:

  * Presence of active electronic implants (e.g., cardiac pacemaker, cochlear implant)
  * Pregnancy (self-reported)
  * History of Epilepsy or seizure disorder
  * Presence of local malignancy (especially near the stimulation site on forearm)
  * Broken skin, wounds, or significant skin conditions on the right forearm (stimulation site)
* Medical/Neurological History:

  * History of significant psychiatric or neurological disease (other than epilepsy, listed above)
  * History of substance dependence
  * Current diagnosis of a chronic pain condition
* Medication Use:

  * Current regular use of prescription analgesic (pain-relief) medication
  * Current regular use of psychoactive medication
* Study-Specific:

  * Self-reported musical anhedonia (inability to derive pleasure from music)
  * Significant hearing impairment preventing clear perception of the music

Ages: 19 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-04-20 (Actual); Study Completion 2025-04-20 (Actual)

PRIMARY OUTCOMES:
Perceived Pain | Time Frame: 40 minutes (duration of time over which each participant is assessed)
  rated on a scale ranging from 1 to 9 (1 = very little, 5 = medium, 9 = very strong)

SECONDARY OUTCOMES:
Emotional state with regard to felt pleasantness | Time Frame: 40 minutes (duration of time over which each participant is assessed)
  rated on a scale ranging from 1 to 9 (1 = very uncomfortable, 5 = medium, 9 = very comfortable)
Emotional state with regard to felt arousal | Time Frame: 40 minutes (duration of time over which each participant is assessed)
  rated on a scale ranging from 1 to 9 (1 = very calm, 5 = medium, 9 = very activated)

OTHER OUTCOMES:
Familiarity with the music excerpt (only during trials with music) | Time Frame: 40 minutes (duration of time over which each participant is assessed)]
  rated on a scale ranging from 1 to 9 (1 = not at all, 5 = partially known, 9 = well known)
Liking ratings for each musical excerpt | Time Frame: 5 min (duration of time over which each participant is assessed)
  rated on a scale ranging from 1 to 9 (1 = strongly disliked, 5 = medium, 9 = strongly liked)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Koelsch, PhD, Principal Investigator — Institute for Biological and Medical Psychology, University of Bergen
Locations (1):
- University of Bergen, Bergen, Norway